CLINICAL TRIAL: NCT03477058
Title: In-Use Test With a Cosmetic Product (WO 3308) for Topical Use to Treat Acute or Chronic Pruritus
Brief Title: In-Use Test With a Cosmetic Product to Treat Pruritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: SIT Skin Investigation and Technology Hamburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPC-17/2016
Record Dates: First submitted 2018-03-15; First posted 2018-03-26 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Pruritus
Keywords: chronic pruritus; acute pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WO 3308 cosmetic product for topical use (Experimental): WO 3308 is used to treat acute or chronic pruritus
  Interventions: Other: WO 3308 cosmetic product for topical use

INTERVENTIONS:
Other: WO 3308 cosmetic product for topical use — Application on the entire body at least once a day over two weeks

SUMMARY:
The aim of the study is to evaluate the cosmetic features of the product WO 3308 by means of a questionnaire in an interview situation after two weeks of product treatment, giving special consideration to the cosmetic performance, efficacy and skin compatibility and with special focus on the reduction of pruritus. Additionally the tolerance will be evaluated by a dermatologist.

ELIGIBILITY:
Inclusion Criteria:

* age: ≥ 18 years
* sex: approx. 25% to 50% male and 50% to 75% female
* with acute pruritus (lasts less than 6 weeks) or chronic pruritus (lasts longer than 6 weeks): max. 50% with acute pruritus and at least 50% with chronic pruritus

Exclusion Criteria:

* any deviation from the above-mentioned criteria
* known incompatibilities to cosmetics and ingredients of cosmetic test products (please see INCI)
* topical medication in the test area within 1 month prior to study start
* systemic medication with antibiotics within 2 weeks prior to starting of the study
* change in the medication with anti-inflammatory agents within 2 weeks prior to starting the study
* systemic medication with immunomodulators (immunsuppressive drugs in the course of a transplantation) and/or chemotherapeutic agents within 4 weeks prior to starting the study
* neurodermatitis (atopic dermatitis)
* pregnancy and period of breastfeeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Cosmetic Features of the Test Product | baseline, two weeks
  Change from baseline for the cosmetic features (spreadability, absorbtion, skin feeling after application, fragrance) of the test product by the means of an interview-based questionnaire
Reduction of Pruritus | baseline, two weeks
  Change from baseline reduction of pruritus at two weeks by the means of an interview-based questionnaire

SECONDARY OUTCOMES:
Tolerance of the Test Product on the skin | baseline, two weeks
  Change from baseline at two weeks by the means of a dermatological and subjective assessment of skin tolerance on arms and legs

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Gust, MD, Study Director — Dermatologist
Locations (1):
- SIT Skin Investigation and Technology Hamburg GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No